CLINICAL TRIAL: NCT07359326
Title: The Effect of Cold Application on Pain, Disease Activity and Quality of Life in Patients With Rheumatoid Arthritis
Brief Title: The Effect of Cold Application in Patients With Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Betül ERTEN, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBU-SBF-BE-01
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cold Application; Pain; Disease Activity; Rheumatoid Arthritis (RA
MeSH Terms: conditions — Pain; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: 2 group with conventional therapy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Application Group (Experimental): Patients will be instructed to apply cold therapy three times daily for 15 minutes each session over a period of three weeks. Patients will report their daily cold application to the researcher via text message. For those unable to provide updates via text, the researcher will follow up daily by phone to monitor adherence to the intervention.
  Interventions: Behavioral: Cold Application
- Control Group (No Intervention): This patient group will undergo follow-up assessment after a three-week period during which no intervention will be administered.

INTERVENTIONS:
Behavioral: Cold Application — Patients will be instructed to apply cold therapy three times daily for 15 minutes each session over a period of three weeks. Patients will report their daily cold application to the researcher via text message. For those unable to provide updates via text, the researcher will follow up daily by phone to monitor adherence to the intervention.
  Arms: Cold Application Group

SUMMARY:
The aim of this thesis is to examine the effects of cold application on pain, disease activity, and quality of life in patients with Rheumatoid Arthritis.

Currently, non-pharmacological interventions, such as cold therapy, are utilized less frequently than pharmacological treatments for the management of pain in inflamed joints. Cold application is anticipated to alleviate pain and consequently enhance patients' quality of life. This study seeks to improve quality of life by reducing pain in patients with Rheumatoid Arthritis. Given its simplicity, ease of application, and low cost, this intervention may be recommended as a pain management strategy both for patients and for nurses working in clinical settings. Furthermore, the study aims to contribute to the existing literature on the subject.

ELIGIBILITY:
Inclusion Criteria

* Having been diagnosed with rheumatoid arthritis at least 6 months ago,
* No problems with speaking, communicating, hearing, or understanding,
* Able to understand and speak Turkish,
* Experiencing pain.

Exclusion Criteria

* Patients who are in remission
* Individuals of foreign nationality
* People with psychiatric or mental illnesses
* Patients who do not consent to participate in the study or who withdraw at any stage of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Rheumatoi Arthritis Disease Activity Index-5 | 3 weeks
  The Rheumatoid Arthritis Disease Activity Index-5 (RADAI-5) is a patient-reported outcome measure designed to assess disease activity in individuals with rheumatoid arthritis

SECONDARY OUTCOMES:
The Short Form Health Survery- SF-36 | 3 weeks
  The Short Form-36 (SF-36) is a widely used generic health-related quality of life (HRQoL) questionnaire designed to assess overall physical and mental well-being. It is a self-administered instrument that evaluates health status across multiple dimensions, making it suitable for clinical practice, research, and population health surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of health sciences Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No